CLINICAL TRIAL: NCT05522309
Title: A Phase I, Open-Label, Multi-Center Dose Finding Study to Investigate the Safety, Pharmacokinetics, and Preliminary Efficacy of FGFR Inhibitor ET0111 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: FGFR Inhibitor ET0111 Monotherapy in Patients With Advanced Solid Tumors
Acronym: FLIGHT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Etern BioPharma (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ET0111-101
Record Dates: First submitted 2022-08-27; First posted 2022-08-31 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Dose Expansion (Experimental): ET0111 will be administered orally once daily in 21 days treatment cycles.
  Interventions: Drug: ET0111

INTERVENTIONS:
Drug: ET0111 — Oral capsules taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 21 days in duration with ET0111 administered, once daily (QD).

SUMMARY:
This is a Phase I, open-label, multi-center, dose-finding study to assess the safety, pharmacokinetics, and preliminary efficacy of ET0111 in patients with advanced solid tumors. It is anticipated that approximately 37 subjects will be enrolled in the dose-escalation phase of the study. ET0111 will be administered orally once daily (QD) in 21-day treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
2. Aged at least 18 years at the time of ICF signature.
3. Histological or cytological confirmation of a solid tumor and have progressed despite standard therapy(ies), or are intolerant to standard therapy (ies), or have a tumor for which no standard therapy(ies) exists. Locally recurrent disease must not be amenable to surgical resection or radiotherapy with curative intent (patients who are considered suitable for surgical or ablative techniques following down-staging with study treatment are not eligible).
4. Estimated life expectancy of minimum of 12 weeks.
5. Patient with solid tumors must have at least 1 lesion, not previously irradiated, that can be accurately measured at pre-dose as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with Computerised Tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at ICF signature.
7. Males and Females of child-bearing potential must agree to use effective contraception from the time ICF signature until 12 weeks after the last dose. Females of childbearing potential include those who are premenopausal and those who are 2 years postmenopausal. Pregnancy tests for female of child-bearing potential must have a negative serum pregnancy test at Screening.

Exclusion Criteria:

1. Have a history and/or current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, vascular system, and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcification..
2. Have current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc.
3. As judged by the investigator, any evidence of significant ophthalmological abnormalities including but not limited to history or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO, retinal macular degeneration, uncontrolled glaucoma, cataract or marked decrease in visual acuity, symptomatic severe dry eye, conjunctivitis, or corneal ulcer.

   Prior bone marrow or organ transplantation
4. Central nervous system metastatic disease, leptomeningeal disease, or metastatic cord compression.
5. Prior therapy with any irreversible FGFR inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) of ET0111 | Approximately 2 years
  MTD based on Number of participants with dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as any toxicity not attributable to the disease or disease-related processes under investigation, which occurs before the end of Cycle 1 (21 days as a cycle)
Recommended Phase 2 Dose (RP2D) | Approximately 2 years
  RP2D may be the same dose level or lower than the determined MTD
Number of participants with adverse events | Approximately 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments

SECONDARY OUTCOMES:
Area under the curve | Approximately 2 years
  Area under the plasma concentration time curve of ET0111
Cmax | Approximately 2 years
  Highest observed plasma concentration of ET0111
Tmax | Approximately 2 years
  Time of highest observed plasma concentration of ET0111
T1/2 | Approximately 2 years
  Half life of ET0111
Objective response rate | Approximately 2 years
  Objective response rate
Duration of response | Approximately 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Disease Control Rate | Approximately 2 years
  DCR is defined as the percentage of patients who achieved remission (PR+CR) and stabilization (SD) after treatment in evaluable cases.
Progression-free survival | Approximately 2 years
  PFS is defined as the time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
Overall survival | Approximately 2 years
  OS is defined as the time between the beginning of randomization and the death of the patient from any cause

OTHER OUTCOMES:
blood phosphorus | Approximately 2 years
  On treatment versus baseline comparison of blood phosphorus
ET0111 metabolites identification | Approximately 2 years
  ET0111 metabolites identify and analysis
NGS test of FGF/FGFR | Approximately 2 years
  Next-generation sequencing (NGS) test will be performed with the tumor tissues or plasma ctDNA collected before ET0111 treatment, to detect FGF/FGFR gene alterations . Detected gene alteration data (including but not limited to mutation, insertion, deletion, amplification, translocation…) will be further analyzed for correlation with the anti-tumor activity of ET0111.

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Principal Investigator — Chinese PLA General Hospital
Locations (5):
- China (5):
  - Beijing Tongren Hospital,CMU, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Zhejiang university school of medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No